CLINICAL TRIAL: NCT02449824
Title: Characterising Early Response to Neoadjuvant Chemotherapy With Quantitative Breast MRI
Brief Title: MRI and Early Decision-making in Chemotherapy for Breast Cancer
Acronym: CHERNAC
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, David Buckley, Professor of Medical Physics, University of Leeds
Other Study IDs: MO15/085
Record Dates: First submitted 2015-05-12; First posted 2015-05-20 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Breast Neoplasms
Keywords: neoadjuvant chemotherapy; magnetic resonance imaging
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumour biopsy samples and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- magnetic resonance imaging: Participants will undergo MRI at baseline, after 1 cycle, 3 cycles and at completion of neoadjuvant chemotherapy.
  Interventions: Other: magnetic resonance imaging

INTERVENTIONS:
Other: magnetic resonance imaging — early MRI
  Other Names: MRI

SUMMARY:
Firstly, the investigators aim to show that breast tumour blood flow, measured as part of a standard MRI examination, decreases at the earliest stage of neoadjuvant chemotherapy in those patients who go on to respond to treatment. Importantly, the investigators will also show that blood flow does not decrease in those patients who fail to respond.

Secondly, the investigators will test whether the decrease in tumour blood flow over the whole course of neoadjuvant chemotherapy can predict the response of the tumour measured at the time of surgery.

DETAILED DESCRIPTION:
i) Background. In a recent pilot study of 18 patients undergoing neoadjuvant chemotherapy (NAC), the investigators demonstrated for the first time that it was feasible to measure breast tumour blood flow (TBF) as part of a standard clinical MRI exam. TBF decreased dramatically in clinical responders and when compared with similar results obtained by others using [15-O] H2O positron emission tomography, the data led the investigators to hypothesise that TBF will decrease after only 1 cycle of NAC in responders. The data also suggested that changes in TBF over the course of NAC might predict pathological response.

ii) Aims. The primary aim is to assess response to first line NAC non-invasively after only 1 cycle of treatment. A secondary aim is to predict pathological response based upon changes measured over the course of NAC.

iii) Techniques and Methodology. The investigators will measure TBF using a novel MRI approach in 40 patients studied before, following 1 cycle, at the mid-point and the end of a fixed course of NAC. The MRI data will be compared with histological and molecular markers, obtained from biopsies at baseline and after 1 cycle of NAC and from specimens obtained during surgery at the end of NAC, to assess mechanisms of response to chemotherapy. In a sub-study of 10 patients imaged twice at baseline the investigators will assess the reproducibility of the TBF measures.

iv) Impact on breast cancer research. These techniques will provide absolute measures of tumour function during therapy which will particularly benefit non-responders to first line NAC allowing clear and objective decisions to be made about possible early changes in their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed large but operable invasive carcinoma of the breast. All molecular subtypes are eligible and incidentally detected small volume metastatic disease is NOT an exclusion criterion.
* Clinical indication for NAC as determined by the Breast Therapeutic MDT.
* Sufficient biopsy material taken at diagnosis to measure the standard molecular markers.
* Participant is willing and able to give informed consent for participation in the study.
* Female, aged 18 years or above.
* Histologically or cytologically confirmed invasive carcinoma of the breast and having received no prior treatment for this.
* Female participants of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study.
* Participant has adequate renal function (estimated glomerular filtration rate ≥ 30 ml/min).
* In the Investigator's opinion, is able and willing to comply with all study requirements.

Exclusion Criteria:

* Previous breast cancer treated with radiotherapy or chemotherapy or recurrent breast cancer.
* Female participant who is pregnant, lactating or planning pregnancy during the course of the study.
* Significant renal impairment (estimated glomerular filtration rate < 30 ml/min).
* Contraindication to MRI.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients aged over 18 years with invasive carcinoma of the breast who, following discussion at the breast multidisciplinary team (MDT) meeting, are to be treated in Leeds using NAC with curative intent will be approached to take part in this study (this includes HER2+ patients receiving trastuzumab); the sample will thus reflect the general population of patients receiving NAC.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change in tumour blood flow between baseline and after 1 cycle of neoadjuvant chemotherapy | 2 weeks
  Cycle 1 length ~ 2 weeks.

SECONDARY OUTCOMES:
Rate of change in tumour blood flow measured at baseline, after 1 cycle, 3 cycles and 6 cycles of NAC & pathological response. | ~18 weeks
  Cycles 1,2 & 3 each of 2 weeks length. Cycles 4, 5 & 6 each of 3 weeks length + short delay before surgery.
Tumour blood flow at baseline, after 1 cycle and after 6 cycles compared with molecular markers measured from biopsy data obtained at baseline and after 1 cycle and measured from surgical specimens taken after 6 cycles. | ~15 weeks
  Cycles 1,2 & 3 each of 2 weeks length. Cycles 4, 5 & 6 each of 3 weeks length.
Within patient coefficient of variation in the measure of blood flow obtained at 2 baseline visits. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David L Buckley, PhD, Principal Investigator — University of Leeds
Locations (1):
- Leeds Teaching Hospitals NHS Trust, St James's University Hospital, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No